CLINICAL TRIAL: NCT06193668
Title: Short-term High-fat Overnutrition Induces Insulin Resistance in White Adipose Tissue
Brief Title: Overfeeding Induced Fat-tissue Stimulation
Acronym: OVID_FASTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OVID-FASTI
Record Dates: First submitted 2022-09-27; First posted 2024-01-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Lipid-induced Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fat overnutrition (Active Comparator): Lipid overnutrition: 40% higher lipid consumption per day than required over three weeks.
  Interventions: Behavioral: High-fat overnutrition
- Normocaloric macronutrient-balanced nutrition (Active Comparator): Normocaloric, macronutrient-balanced nutrition per day over three weeks
  Interventions: Behavioral: Normocaloric macronutrient-balanced nutrition

INTERVENTIONS:
Behavioral: High-fat overnutrition — Overnutrition: 40% higher lipid consumption per day than required
  Arms: High-fat overnutrition
Behavioral: Normocaloric macronutrient-balanced nutrition — Normocaloric, macronutrient-balanced nutrition:
  Calories requirement for weight maintenance [(kcal/d) 55% carbohydrates, 15% proteins, 30% fat]
  Arms: Normocaloric macronutrient-balanced nutrition

SUMMARY:
Type 2 diabetes is the most common metabolic disease worldwide, characterized by hyperglycemia, decreased whole body insulin sensitivity, and white adipose tissue (WAT) dysfunction. A key factor in its development is chronic overnutrition, usually with a high-fat diet (HFD), leading to disturbances of glucose and lipid metabolism. However, the mechanism of short-term HFD-induced tissue-specific insulin resistance remains poorly understood. This project aims to further unravel the underlying mechanisms of short-term HFD overnutrition-mediated WAT insulin resistance. The model described here corresponds to a randomized, single- blinded parallel-grouped trial, consisting of two interventions: a macronutrient-balanced diet and or a hypercaloric diet over three weeks in order to investigate differences in interorgan fatty acid and glucose metabolism between the studied groups. Based on recent studies, the hypothesis is that 21-day hypercaloric HFD induces WAT insulin resistance via a diacylglycerol, novel protein kinase C-insulin receptor signaling model in both fasting and insulin-stimulated states.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* BMI < 29 kg/m2
* Sport inactive (<1x /week)
* Capacity to consent

Exclusion Criteria:

* Diabetes mellitus disease
* Acute coronary heart syndrome (myocardial infarction, unstable angina pectoris, stroke or transient ischemic attack in the last 3 months before study participation)
* Acute infectious disease
* Taking blood glucose-lowering drugs
* Diseases or drugs affecting the immune system and allergies to drugs used in the study
* Drugs with potential metabolic effects
* Chronic liver disease (hepatitis, gallbladder disease, elevated liver enzymes (ALT > 300 U/L))
* Chronic inflammatory bowel diseases
* Rheumatic diseases
* Hyper- or hypothyroidism of the thyroid gland
* Renal insufficiency, administration of iodine-containing contrast media in the last 2 days
* Chronic lung diseases
* cancerous diseases
* Addictive diseases, psychiatric diseases
* Pregnancy, breastfeeding
* Shift workers
* Anemia (Hb <12 g/dl)
* Disorders of hemostasis
* Regular use of antithrombotic drugs
* Alcohol consumption, smoking
* Conditions that do not permit an MRI examination

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Whole-body insulin sensitivity and WAT insulin sensitivity | 3 weeks intervention period each
  Hyperinsulinemica-euglycemia clamp tests with deuterated glucose to measure fasting and insulin-stimulated whole-body insulin sensitivity and measurement of the index ADIPO-IR (fasting insulin x free fatty acid concentration) before and after dietary intervention period.

SECONDARY OUTCOMES:
WAT insulin signaling pathways | 3 weeks intervention time
  Adipose tissue biopsies are planned to be taken during the fasting and insulin-stimulated state before and after the dietary intervention period. DAG and ceramide subcellular fractionation assay is planned to be performed. Expressionanalyses for activation /membrane translocation of novel and atypical protein kinase C isoforms will be done. Determination of the degree of phosphorylation of various components of the insulin pathway via Western blot are planned.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Study Director — German Diabetes Center
Locations (1):
- Georgia Xourafa, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No